CLINICAL TRIAL: NCT03657290
Title: A Randomized, Open-Label, Single-Dose, Three-Period Six-Sequence Crossover Study in Healthy Adults to Assess Bioequivalence Between Test and Reference Vadadustat 450 mg and 150 mg Tablets and to Determine Food Effect on the 450 mg Vadadustat Tablet.
Brief Title: A Study in Evaluating Bioequivalence of Test and Reference Vadadustat 450 MG and 150 MG Tablets and to Determine Food Effect on the 450 MG Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0028
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Vadadustat; healthy volunteers; bioequivalence; pharmacokinetics
MeSH Terms: interventions — vadadustat

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, single-dose, three-period, six- sequence crossover study in healthy adults. A total of 54 eligible subjects will be randomized to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA). Refer to Treatment Sequences below. Each sequence is comprised of 3 treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): vadadustat 3 X 150 mg Tablets in fasted subjects
  Interventions: Drug: vadadustat
- Treatment B (Active Comparator): Vadadustat 1 X 450 mg Tablets in fasted subjects
  Interventions: Drug: vadadustat
- Treatment C (Active Comparator): vadadustat 1 X 450 mg Tablets in fed subjects
  Interventions: Drug: vadadustat

INTERVENTIONS:
Drug: vadadustat — Vadadustat Tablets
  Other Names: AKB-6548

SUMMARY:
This is a healthy volunteers study to assess the bioequivalence of vadadustat 450 mg tablets (Test A) compared to three 150mg tablets (Reference B). The study will also assess the effect of food on the bioavailability of vadadustat 450 mg tablet.

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose, three-period crossover study in healthy adults to assess the bioequivalence of 3 X 150 mg vadadustat tablets (Test) compared to a single 450 mg vadadustat tablet (reference). Blood samples for vadadustat PK will be collected at pre-dose (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, 32, 40, and 48 hours post-dose. The study will also assess the effect of food on vadadustat bioavailability by evaluating the pharmacokinetics of the 450 mg tablet in fed and fasted subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between ≥18 years and ≤55 years of age
* Healthy subjects per Investigator judgment as documented by the medical history, physical examination, vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and general observations.
* Have a body weight ≥50 kg and body mass index (BMI) ≥18.5 kg/m2 to 29.5 kg/m2 inclusive
* Understands the procedures, provides ICF and willing to comply with study requirements
* Willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease.
* History of cancer (except non- melanoma skin cancer) or history of chemotherapy use.
* Any surgical or medical condition or history that may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to gastric bypass surgery or gastric or duodenal ulcers.
* History of severe allergic or anaphylactic reactions. Chronic daily medication use.
* History of drug abuse Excessive alcohol consumption.
* Smoking and the use of nicotine-containing products
* Consumption of grapefruit or grapefruit juice, pomelo, star fruit, Seville or Moro (blood) orange, or their associated products
* Participation in another clinical trial or exposure to any investigational agent.
* Donation of blood or significant blood loss or plasma donation.
* Any condition that would interfere with the ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the patient at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Bioequivalence - Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) | Baseline visit, 48 hours
Bioequivalence - Area under plasma concentration-time curve from 0 to infinity (AUCinf) | Baseline visit, 48 hours
Bioequivalence - Area under plasma concentration-time curve from 0 to last sampling point (AUCall) | Baseline visit, 48 hours
Bioequivalence - Observed Maximum concentration (Cmax) | Baseline visit, 48 hours
Measure Food Effect - Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) | Baseline visit, 48 hours
Measure Food Effect - 2. Area under plasma concentration-time curve from 0 to infinity (AUCinf) | Baseline visit, 48 hours
Measure Food Effect - 2.3. Observed Maximum concentration (Cmax) | Baseline visit, 48 hours

SECONDARY OUTCOMES:
Time to reach Cmax | Baseline visit, 48 hours
Time to reach Tmax | Baseline visit, 48 hours
Mean residence time (MRT) | Baseline visit, 48 hours
Elimination rate constant (Kel) | Baseline visit, 48 hours
Apparent total body clearance (CL/F) | Baseline visit, 48 hours
Apparent volume of distribution (Vd/F) | Baseline visit, 48 hours
Terminal half-life (t1/2) | Baseline visit, 48 hours
Percentage of extrapolated area under the curve from time t to infinity (AUCextrap or Residual Area) | Baseline visit, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- Paraxel International, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided